CLINICAL TRIAL: NCT01616186
Title: A Randomized Non-Comparative Multicenter Phase II Study of Everolimus/Sorafenib or Sunitinib in Patients With Metastatic Renal Cell Carcinoma (RCC)
Brief Title: Everolimus/Sorafenib or Sunitinib in Patients With Metastatic Renal Cell Carcinoma (RCC)
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Andrea Harzstark (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor-Investigator, Andrea Harzstark, Clinical Professor, UCSF Helen Diller Cancer Center, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSF CC# 12521
Record Dates: First submitted 2012-06-04; First posted 2012-06-11 (Estimated); Last update posted 2013-04-08 (Estimated); Status verified 2013-04

CONDITIONS: Locally Metastatic Malignant Neoplasm
Keywords: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Everolimus; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Everolimus/Sorafenib (Experimental): Patients will be stratified by current smoking status (smoker: yes or no0, for each smoking stratum patients will be randomized in a 2:1 ratio
  Interventions: Drug: Everolimus and sorafenib
- Sunitinib (Active Comparator): * Sunitinib is the concurrent control group
  * Patients will be stratified by current smoking status (smoker: yes or no), for each smoking stratum patients will be randomized in a 2:1 ratio
  Interventions: Drug: Sunitinib monotherapy

INTERVENTIONS:
Drug: Everolimus and sorafenib — * Starting doses: everolimus 5 mg daily and sorafenib 400 mg BID - taken fasting, no food 1 hour before or 2 hours after dosing
  * Everolimus and sorafenib are dosed continuously
  (Note: everolimus and sorafenib are typically dosed in 28 day cycles, and sunitinib is typically dosed in 42 day cycles; for the purposes of this protocol to keep timing consistent, a cycle will be defined as 42 days of therapy)
  Arms: Everolimus/Sorafenib
Drug: Sunitinib monotherapy — Starting dose: sunitinib 50 mg daily 4 weeks on, 2 weeks off - taken fasting, no food 1 hour before or 2 hours after dosing
  (Note: sunitinib is typically dosed in 42 day cycles described above: 28 days treatment, 14 days off. For the purposes of this protocol, to keep timing consistent, a cycle will be defined as 42 days of therapy)
  Arms: Sunitinib

SUMMARY:
This is a phase II trial that follows the completion of the phase I UCSF trial of everolimus and sorafenib for Renal Cell Carcinoma (RCC). This trial will be for patients who have not had treatment for RCC before. This trial will have 2/3 patients getting everolimus/sorafenib treatment and 1/3 getting sunitinib, an FDA approved RCC drug. All three drugs are approved for advanced RCC when used individually, the combination of everolimus and sorafenib for RCC is not approved by the FDA.

DETAILED DESCRIPTION:
In the phase I study of the combination of everolimus and sorafenib, clinical benefit was observed in patients with no prior systemic therapy. There was no evidence of pharmacokinetic interaction and acceptable toxicity at a dosage of sorafenib of 400 mg twice daily (BID) and everolimus 5 mg daily. Based on these data and the need for more effective front-line therapy for renal cell carcinoma, the plan is to investigate this regimen in patients who have not undergone prior therapy. A sunitinib arm is being included as a concurrent reference to help provide a guideline of an activity level and toxicity that would be meaningful to move forward to a phase III study. Therefore, this study is designed as a non-comparative investigation and patients will be randomized in a 2:1 ratio to everolimus/sorafenib or to sunitinib, respectively.

ELIGIBILITY:
INCLUSION CRITERIA

1. Histologically- or cytologically-confirmed renal cell carcinoma, which is unresectable or metastatic and of any of the following histologies: clear cell, papillary, chromophobic, oncocytic, unclassified, or mixed. A component of clear cell histology must be present. Tumors with pure collecting duct histology are not eligible.
2. Cytoreductive nephrectomy is allowed but not required
3. Evidence of RECIST-defined measurable disease (lesions that can be accurately measured in at least one dimension with the longest diameter ≥ 20mm using conventional techniques or ≥ 10 mm with spiral CT scan)
4. Male or female at least 18 years old

   1. Female patients must be either surgically sterile or postmenopausal, or if of childbearing potential must have a negative pregnancy test (serum or urine) prior to enrollment and agree to use effective barrier contraception during the period of therapy, and for 3 months after the end of treatment/end of participation in the study. Oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study.
   2. Male patients must be surgically sterile or must agree to use effective contraception during the period of therapy, and for 3 months after the end of treatment/end of participation in the study.
   3. The definition of effective contraception will be based on the judgment of the investigator.
5. ECOG performance status 0-1
6. Adequate bone marrow function:

   1. ANC ≥ 1500/uL
   2. platelet count ≥ 100,000/uL
   3. hemoglobin ≥ 9.0 g/dL
7. Adequate hepatic function:

   1. Total bilirubin ≤ 1.5 X ULN
   2. AST (SGOT) ≤ 2.5 X ULN
   3. ALT (SGPT) ≤ 2.5 X ULN
8. Adequate renal function as determined by either:

   1. Calculated or measured creatinine clearance ≥ 40 mL/min (for calculated creatinine clearance, Cockroft-Gault equation will be used)

      Modified Cockcroft-Gault formula:

      ((140 - age (yrs)) x (actual weight(kg))) / (72 x serum creatinine(mg/dl))

      * Multiply by another factor of 0.85 if female
   2. Serum creatinine ≤ 1.5 X ULN
9. Able to swallow oral medications
10. Total fasting serum cholesterol ≤ 300 mg/dL
11. Resolution of any pre-existing toxicity from prior therapy to NCI CTCAE V3.0 ≤ grade 1 (with the exception of hypertension, hypothyroidism)
12. Signed and dated informed consent document
13. Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedures.
14. More than 28 days since any prior therapy, including investigational agents and surgical procedures.

EXCLUSION CRITERIA

1. Collecting duct renal cell carcinoma is excluded. Transitional cell carcinoma of the renal pelvis is excluded.
2. Prior systemic regimens for renal cell carcinoma (neoadjuvant therapy is acceptable as long as it did not include sunitinib, sorafenib, everolimus, or temsirolimus). A prior therapy which was started and stopped after no more than four weeks of therapy will not constitute a prior systemic regimen.
3. Prior surgery, radiation therapy, or systemic therapy for renal cell carcinoma within 4 weeks of starting study treatment.
4. History of or known brain metastasis, spinal cord compression, or carcinomatous meningitis, or new evidence of brain or leptomeningeal disease on screening CT or MRI scan (evaluation for CNS disease is required to be performed for eligibility).
5. Any of the following within 6 months prior to study drug administration: myocardial infarction, unstable or severe angina, coronary or peripheral artery bypass graft, NYHA functional Class II, III, IV congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
6. Ejection fraction lower than institutional lower limit of normal by echocardiogram or MUGA.
7. Hypertension that is unable to be controlled with medications to a blood pressure of ≤ 150/90.
8. Hypothyroidism that is unable to be controlled with medications such that FT4 is outside of normal limits.
9. QTc prolongation (QTc interval ≥ 480 msecs) or any other clinically significant ECG abnormalities.
10. Known human immunodeficiency virus (HIV) or acquired immune deficiency syndrome (AIDS)-related illness (because of the immunosuppressive effects of therapy). Testing for HIV in the absence of a history or symptoms is not required.
11. Hepatitis B or C (because of the risk of reactivation). The following serologies are acceptable for enrollment: HBsAg-/anti-HBc-/anti-HBs-; HBsAg-/anti-HBc+/anti-HBs+; HBsAg-/anti-HBc-/anti-HBs+. The following serologies are not acceptable for enrollment: HBsAg+/anti-HBc+(IgM+/-)/anti-HBs-. If the following serologies are obtained, additional testing will be required to ascertain the patient's hepatitis B status: HBsAg-/anti-HBc+/anti-HBs-.
12. "Currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered to have a less than 30% risk of relapse.
13. Current treatment on another clinical trial.
14. Pregnant or breastfeeding.
15. Chronic treatment with systemic steroids or other immunosuppressive agent.
16. On oral vitamin K antagonist medication (except low dose warfarin) (other anticoagulants are allowed).
17. History of malabsorption syndrome, disease significantly affecting gastrointestinal function or major resection of stomach or small bowel that could interfere with absorption, distribution, metabolism, or excretion of study drugs.
18. Any serious and/or unstable pre-existing medical, psychiatric, or other condition (including lab abnormalities) that could interfere with subject safety or obtaining informed consent. Examples of such include uncontrolled diabetes as defined by fasting serum glucose >1.5 x ULN (Note: optimal glycemic control should be achieved before starting trial therapy), nonhealing wound, severe infection, severe malnutrition, ventricular arrhythmias, active ischemic heart disease, chronic liver or renal disease, or active upper GI tract ulceration.
19. Patients should not receive immunization with attenuated live vaccines within one week of study entry or during study period. Close contact with those who have received attenuated live vaccines should be avoided during treatment with everolimus. Examples of live vaccines include intranasal influenza, measles, mumps, rubella, oral polio, BCG, yellow fever, varicella and TY21a typhoid vaccines.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Objective response | 12-18 weeks
  Computerized Tomography Scans (CT) done at Screening and every 2 cycles
  * For Partial Response (PR) or Complete Response (CR), changes in tumor measurements must be confirmed by repeat studies no less than 4 weeks after the criteria for response are first met (RECIST 1.1 criteria)
  * For Stable Disease (SD), follow-up measurements must have met the SD criteria at least once after study entry at a minimum of 12 weeks after study entry

SECONDARY OUTCOMES:
Safety: combination of everolimus and sorafenib | 12-18 weeks
  Safety/Adverse Event (AE) assessments done on Day 1, 21, 42 during Cycle 1 & Day 28 of all subsuquent cycles; assessments include Eastern Oncology Group Conference (ECOG) Performance scale, physical/history, hematology & chemistry labs; other safety data (e.g. Electrocardiogram [ECG], Multigated Acquisition Scan [MUGA], etc.) will be considered as appropriate
Progression-free Survival (PFS) | 12-18 weeks
  - PFS will be measured (using RECIST 1.1 criteria) from the start of protocol therapy until the date of the first occurrence of recurrent or progressive disease or death
Time-to-Progression (TTP) | 12-18 weeks
  - TTP will be measured from the start of protocol therapy until first date that recurrent or progressive disease is documented
Clinical Benefit rate | 12-18 weeks
  Clinical benefit (defined as objective response+stable disease) will be summarized for each treatment arm by the proportion of patients achieving this outcome with 95% confidence intervals

CONTACTS AND LOCATIONS:
Overall Officials: Andrea Harzstark, MD, Study Chair — University of California, San Francisco